CLINICAL TRIAL: NCT01568320
Title: Use of the Zenith® Dissection Endovascular System in the Treatment of Patients With Acute, Complicated Type B Aortic Dissection
Brief Title: Zenith® Dissection Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-007
Expanded Access: NCT02464943 (Approved for marketing)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Aortic Dissection
Keywords: Aorta; Thoracic; Aortic dissection; Rupture; Type B; DeBakey type III; Endovascular
MeSH Terms: conditions — Aortic Dissection; Rupture | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Endovascular (Experimental): Endovascular Treatment (Zenith)
  Interventions: Device: Endovascular Treatment (Zenith)

INTERVENTIONS:
Device: Endovascular Treatment (Zenith) — Instead of making a large incision in the chest, the physician makes a small incision near each hip to insert, and guides the study device(s) into place in the aorta.
  Other Names: Endovascular graft; Endovascular stent; Stent-graft

SUMMARY:
The Zenith® Dissection Clinical Trial is a clinical trial approved by US FDA to study the safety and effectiveness of the Zenith® Dissection Endovascular System in the treatment of acute, complicate Type B aortic dissection.

ELIGIBILITY:
Exclusion Criteria:

1. Age < 18 years;
2. Other medical condition (e.g., cancer, congestive heart failure) that may cause the patient to be non-compliant with the Clinical Investigation Plan, confound the results, or is associated with limited life expectancy (i.e., less than 2 years);
3. Pregnant, breast-feeding, or planning on becoming pregnant within 60 months;
4. Unwilling or unable to comply with the follow-up schedule;
5. Inability or refusal to give informed consent;
6. Simultaneously participating in another investigative device or drug study. (The patient must have completed the primary endpoint of any previous study at least 30 days prior to enrollment in this study.);
7. Additional medical restrictions as specified in the Clinical Investigation Plan; or
8. Additional anatomical restrictions as specified in the Clinical Investigation Plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lombardi, MD, Principal Investigator — The Cooper Health System
Locations (24):
- United States (23):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Indiana Heart Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York University Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - Scott and White Hospital, Temple, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Sentara Vascular Specialists, Norfolk, Virginia
  - University of Washington-Harborview Medical Center, Seattle, Washington
- Jikei University School of Medicine, Tokyo, Japan

REFERENCES:
- [Derived] Lombardi JV, Gleason TG, Panneton JM, Starnes BW, Dake MD, Haulon S, Mossop PJ, Seale MM, Zhou Q; STABLE II Investigators. STABLE II clinical trial on endovascular treatment of acute, complicated type B aortic dissection with a composite device design. J Vasc Surg. 2020 Apr;71(4):1077-1087.e2. doi: 10.1016/j.jvs.2019.06.189. Epub 2019 Aug 30. PMID 31477479

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endovascular
Started | 73
5-Year | 36 (Patients eligible for Follow-up at 5 year)
Completed | 32
Not Completed | 41
Not completed — Death | 20
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 10
Not completed — Conversion to open repair | 1
Not completed — Patient fell outside of the consented window, data outside of the consented 5-year was not collected | 1

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From Major Adverse Events
Description: Primary safety : Major adverse events include: myocardial infarction, chronic renal insufficiency/chronic renal failure requiring dialysis, bowel ischemia, stroke, paraplegia or paraparesis, and prolonged ventilator support
Time Frame: 30 days
Population: In accordance with a revised data analysis plan approved under the IDE , 6 patients were excluded from the hypothesis testing due to meeting certain medical exclusion criteria (i.e., patients who were ASA class V or who were without confirmed absence of bowel necrosis at the time of enrollment).Additional information/reference why no analysis was performed for 6 patients is listed in the CIP in section 7.1
Measure: Number; unit: participants
Arm/Group | Endovascular
Number analyzed (Participants) | 67
participants | 48
Statistical Analysis 1: Comparison: Endovascular; Test type: Superiority or Other; Freedom from Major adverse events (%) = 71.6, 95% CI 2-sided [59 to 82] — Clopper-Pearson (Exact) Method

2. Primary Outcome: Survival Rate at 30 Days
Description: Primary effectiveness endpoint is freedom from all cause mortality at 30 days
Time Frame: 30 days
Population: In accordance with a revised data analysis plan approved under the IDE , 6 patients were excluded from the hypothesis testing due to meeting certain medical exclusion criteria (i.e., patients who were ASA class V or who were without confirmed absence of bowel necrosis at the time of enrollment). Additional information/reference why no analysis was performed for 6 patients is listed in the CIP in section 7.1
Measure: Number; unit: participants
Arm/Group | Endovascular
Number analyzed (Participants) | 67
participants | 64
Statistical Analysis 1: Comparison: Endovascular; Test type: Superiority or Other; Survival rate (%) = 95.5, 95% CI 2-sided [87 to 99] — Clopper-Pearson (Exact) Method

ADVERSE EVENTS:
Time Frame: 5-Year
Arm/Group | Endovascular
All-Cause Mortality (participants affected / at risk) | 20/73
Serious Adverse Events (participants affected / at risk) | 63/73
Other Adverse Events (participants affected / at risk) | 40/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular (N=73)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 4 (4)
Arrhythmia (Cardiac disorders) | 4 (4)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 3 (3)
Cataract (Eye disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1)
Gastoroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastric volvulus (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine ulcer (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Mouth swelling (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 5 (5)
Mucosal inflammation (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 3 (3)
Nodule (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Stent-graft endoleak (General disorders) | 3 (4)
Swelling (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bacillus infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Sepsis (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Vascular access site infection (Infections and infestations) | 2 (2)
Vascular device infection (Infections and infestations) | 1 (1)
Device use error (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (2)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (3)
Blood creatinine increased (Investigations) | 2 (2)
White blood cell count increased (Investigations) | 1 (1)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Arthraglia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Lethargy (Nervous system disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Paraparesis (Nervous system disorders) | 2 (2)
Paraplegia (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (4)
Device lead damage (Product Issues) | 1 (1)
Stent malfunction (Product Issues) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (3)
Renal failure (Renal and urinary disorders) | 7 (8)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Enterostomy (Surgical and medical procedures) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1)
Mechanical ventilation (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 6 (6)
Aortic dissection (Vascular disorders) | 6 (8)
Aortic rupture (Vascular disorders) | 2 (2)
Arterial thrombosis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypertensive urgency (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Iliac artery dissection (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 2 (2)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 2 (2)
Malignant hypertension (Vascular disorders) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 2 (2)
Subclavian steal syndrome (Vascular disorders) | 1 (1)
Thrombus (Vascular disorders) | 1 (1)
Vascular dissection (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular (N=73)
Anaemia (Blood and lymphatic system disorders) | 9 (10)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5)
Arrhythmia (Cardiac disorders) | 8 (11)
Chest pain (General disorders) | 6 (8)
Urinary tract infection (Infections and infestations) | 11 (14)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Headache (Nervous system disorders) | 4 (5)
Urinary retention (Renal and urinary disorders) | 7 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Hypertension (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT01568320/Prot_SAP_000.pdf